CLINICAL TRIAL: NCT04299282
Title: A Prospective, Randomized, Single-Center Study Evaluating CanGaroo in Low BMI Patients Undergoing Pacemaker, ICD, or S-ICD Implantation
Brief Title: CIED Implantation in Low BMI Patients
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Postponed due to COVID-19 pandemic
Sponsor: Elutia Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CPR-2205
Record Dates: First submitted 2020-03-05; First posted 2020-03-06 (Actual); Last update posted 2025-05-16 (Actual); Status verified 2025-05

CONDITIONS: Heart Diseases; Cardiac Disease
Keywords: CIED, Pacemaker, ICD, S-ICD
MeSH Terms: conditions — Heart Diseases

STUDY DESIGN:
Intervention Model Description: Randomized 1:1 for 10 in the treatment group and 10 in the control group, shall be enrolled
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- CanGaroo (Active Comparator): The treatment group will receive a CanGaroo envelope with implantation of a CIED
  Interventions: Device: CanGaroo
- No CanGaroo (No Intervention): The control group will not receive a CanGaroo envelope with implantation of a CIED

INTERVENTIONS:
Device: CanGaroo — CIED ECM envelope
  Arms: CanGaroo

SUMMARY:
The primary objective is to demonstrate a better degree of healing at the incision site and a decrease in erosion with CanGaroo compared to control patients (no envelope, CIED alone).

DETAILED DESCRIPTION:
A single-center, prospective, randomized, post-market study of patients undergoing implantation of a pacemaker, ICD, or S-ICD with or without CanGaroo using the same hydration solution. Twenty patients, randomized 1:1 for 10 in the treatment group and 10 in the control group, shall be enrolled. Follow-up visits include post-op and 3-months following the implantation procedure.

ELIGIBILITY:
Inclusion Criteria:

* BMI of less than 23.
* Already scheduled for or a clinical decision made to have one of the following qualifying CIED implant procedures using a device cleared by the U.S. FDA:

  * De novo pacemaker, ICD, or S-ICD;
  * Upgrade or change out of existing CIED to a pacemaker, ICD, or S-ICD
* Clinically stable and able to tolerate procedure.
* Be able and willing to return for follow-up care through the 3-month visit.
* Must possess the ability to provide informed consent.

Exclusion Criteria:

* Patients with a known sensitivity to porcine material.
* Participation in another clinical study.
* Active infection. Clinical diagnosis of an active infection at the time of CIED implant (CIED infection, pneumonia, UTI, endovascular, cellulitis, bacteremia, or other major systemic infection).
* Female patient who is pregnant, or planning to become pregnant during the length of the study.
* Prior history of a CIED infection, other prosthetic device infection, or endovascular infection, including endocarditis in the past 12 months.
* Life expectancy of less than 3 months.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-06 (Estimated); Primary Completion 2021-12 (Estimated); Study Completion 2022-03 (Estimated)

PRIMARY OUTCOMES:
Healing at incision site | 3 months post CIED implantation
  Improved incision site healing for the CanGaroo group

SECONDARY OUTCOMES:
QOL Survey | 3 months post CIED implantation
  Patient assessment via Quality of Life Survey
Vascular Tissue Layer | 3 months post CIED implantation
  Ultrasound measurement of vascular tissue layer
Skin Fold Test | 3 months post CIED implantation
  Skin fold test measurement for tissue thickness

CONTACTS AND LOCATIONS:
Overall Officials: Jerry Riebman, MD, MA, Study Director — Elutia Inc.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Sponsor website — http://www.aziyo.com